CLINICAL TRIAL: NCT00251784
Title: A Double-Blind, Randomised, Placebo Controlled Healthy Volunteer Study to Investigate the Nature and Origin of the Disturbance of Vision Induced by Single Oral Doses of Sildenafil
Brief Title: Healthy Volunteer Study of Sildenafil Effects Upon Vision
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cambridge (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Educational/Counseling/Training
Other Study IDs: LREC 98/297
Record Dates: First submitted 2005-11-09; First posted 2005-11-10 (Estimated); Last update posted 2005-11-10 (Estimated); Status verified 2003-12

CONDITIONS: Blindness
MeSH Terms: conditions — Blindness | interventions — Sildenafil Citrate

INTERVENTIONS:
Drug: Sildenafil

SUMMARY:
Patients sometimes report subjective visual effects when taking sildenafil. Our study set out to measure these in a controlled setting. Subjects were asked to detect patterns presented on a monitor screen.

ELIGIBILITY:
Inclusion Criteria: male -

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2002-02; Study Completion 2003-06

CONTACTS AND LOCATIONS:
Overall Officials: Morris J Brown, MD, Principal Investigator — University of Cambridge; John Mollon, FRS, Study Director — University of Cambridge